CLINICAL TRIAL: NCT01599507
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Sequential Group, Dose Ranging Safety and Efficacy Study of FG 4592 in Non-dialysis Chronic Kidney Disease (CKD) Subjects With Anemia
Brief Title: Study of FG-4592 in Subjects With Chronic Kidney Disease in China
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FGCL-4592-047
Record Dates: First submitted 2012-05-11; First posted 2012-05-16 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Anemia in Chronic Kidney Disease
Keywords: Anemia; Renal
MeSH Terms: conditions — Anemia | interventions — roxadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FG-4592 (Experimental): Active Drug
  Interventions: Drug: FG-4592
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FG-4592 — TIW dosing, capsule
  Arms: FG-4592
Drug: Placebo — TIW dosing, capsule
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate efficacy and safety of FG-4592 in the correction of anemia in non-dialysis chronic kidney disease patients.

DETAILED DESCRIPTION:
Dose ranging study with two consecutive dose escalation cohorts. The study objective is to demonstrate that FG-4592 is effective in the correction of anemia in chronic kidney disease patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years
2. Subject has voluntarily signed and dated an informed consent form
3. Chronic Kidney Disease, not receiving dialysis
4. Hemoglobin (Hb) values in 4 screening visits and the mean Hb must be <10g/dL
5. Aminotransferase levels (alanine aminotransferase [ALT], aspartate aminotransferase [AST]) and total bilirubin must be ≤ upper limit of normal (ULN) during the screening period
6. Serum alkaline phosphatase (ALP) ≤2x ULN during screening period. Subjects with serum ALP values between 1 x and 2 x ULN may be included only if bone-specific ALP (BSAP) is also elevated > ULN
7. Total bilirubin values must be ≤ULN during screening period
8. Serum folate and vitamin B12 levels above the lower limit of normal (LLN)
9. Body weight: 40 to 100 kg (dry weight) inclusive
10. Body mass index (BMI): 16 to 38 kg/m2 inclusive

Exclusion Criteria:

1. Received any erythropoiesis-stimulating agent (ESA) other than epoetin alfa within 12 weeks prior to Day 1
2. Any clinically significant infection or evidence of an underlying infection such as a white blood cell count (WBC) > ULN during screening on two separate occasions,
3. Positive for any of the following: human immunodeficiency virus (HIV); hepatitis B surface antigen (HBsAg); anti-hepatitis C virus antibody (anti-HCV Ab)
4. History of chronic liver disease
5. New York Heart Association Class III or IV congestive heart failure
6. Chronic inflammatory disease other than glomerulonephritis that could impact erythropoiesis (e.g., systemic lupus erythematosis, rheumatoid arthritis, celiac disease) even if it is currently in remission
7. Active or chronic gastrointestinal bleeding, or a known coagulation disorder
8. Hemoglobinopathy (e.g., homozygous sickle-cell disease, thalassemia of all types, etc.)
9. Hematological disorders, including myelodysplastic syndrome, multiple myeloma, or pure red cell aplasia
10. History of hemosiderosis, hemochromatosis, polycystic kidney disease, or anephric
11. Active hemolysis or diagnosis of hemolytic syndrome
12. Known bone marrow fibrosis
13. Uncontrolled or symptomatic secondary hyperparathyroidism (PTH>600ng/L)
14. Any prior organ transplantation
15. Drug-treated gastroparesis, short-bowel syndrome, or any other gastrointestinal condition that may lead to reduced absorption of study drug
16. Serum albumin <3 g/dL
17. History of alcohol or drug abuse; or a positive drug screen for a substance that has not been prescribed for the subject
18. Prior treatment with FG-4592
19. Use of an investigational medication or treatment, or carryover effect of an investigational treatment expected, during the screening visit, treatment and follow-up period.
20. Use of traditional Chinese medicines (TCM) during the screening visit to Day 1 or plans to use TCM during the study unless approved in advance by the Medical Monitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Maximum change in hemoglobin by Week 9 from baseline | Week 9

SECONDARY OUTCOMES:
Proportion of subjects achieving a target Hb level ≥11 g/dL by Weeks 5,6,7,8 and 9. | Week 9
Proportion of subjects with a Hb increase from baseline ≥1.0 g/dL. | Week 9

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital, Chengdu
  - First affiliated hospital of Dalian medical university, Dalian
  - First Affiliated Hospital, Sun Yat-Sen University, Guangzhou
  - Zhejiang University No 1. Hospital, Hangzhou
  - Chang Zheng Hospital, Shanghai
  - Huashan Hospital, Shanghai
  - Renji Hospital, Shanghai
  - RuiJin Hospital, Shanghai
  - XinHua Hospital, Shanghai
  - Shenzhen People's Hospital, Shenzhen

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278